CLINICAL TRIAL: NCT00645255
Title: A Multicenter, Double-Blind, Placebo-Controlled, Parallel Group Study to Examine the Longer-Term Efficacy and Safety of Meridia (Sibutramine Hydrochloride) in Obese Subjects
Brief Title: Study to Examine the Longer-Term Efficacy and Safety of Sibutramine Hydrochloride in Obese Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Peter Bacher, MD, PhD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB118
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Single-blind Placebo Run-in with behavioral intervention called Health Management Resources Maintenance Program which provided weekly classes for 12 months with meal replacement
  Interventions: Drug: placebo
- 2 (Placebo Comparator): Double-blind Treatment with behavioral intervention called Health Management Resources Maintenance Program which provided weekly classes for 12 months with meal replacement
  Interventions: Drug: sibutramine or placebo

INTERVENTIONS:
Drug: placebo — placebo one capsule daily
  Arms: 1
Drug: sibutramine or placebo — one capsule daily
  Other Names: ABT-911; Meridia; sibutramine
  Arms: 2

SUMMARY:
The study was designed to evaluate the long term efficacy and safety of Meridia 15 mg daily in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be able to communicate meaningfully with the investigator, be legally competent, provide written informed consent, and follow a specified diet and exercise program.
* Female subjects must be nonlactating and must either be a) at least one year postmenopausal; or b) surgically sterilized by bilateral tubal ligation, bilateral oophorectomy or hysterectomy; or c) using adequate contraceptive precautions (i.e., oral contraceptives, approved hormonal implant, intrauterine device, diaphragm with spermicide, condom with spermicide).
* A serum pregnancy test, which must be negative, is required of all females except those who are surgically sterile or postmenopausal.
* The subject must be at least 18 years old.
* The subject must have a systolic blood pressure <=140 mmHg, a diastolic blood pressure<=90 mmHg, and a pulse rate <=95 beats per minute (see Section VI.I.). Treated hypertensives are allowed in the study.
* The subject must have been enrolled in a nonpharmacologic weight loss program with documented weight loss of >=10 kg maintained for at least 6 months, have gained back <50% of their peak lost weight (while currently maintaining a weight loss of >=10 kg), and be stabilized on a weight-maintaining diet for at least 1 month prior to screening.
* The subject's body mass index (BMI) must be >=27 kg/m2 and <=40 kg/mg2, rounded to the nearest whole unit, and must have been >=30 kg/m2 prior to initiation of the nonpharmacological weight loss program prior to screening.
* The subject must have lived in the immediate geographic area for at least 2 years prior to screening.
* If the subject is on chronic medication, the dose must have been constant for at least two months prior to screening.

Exclusion Criteria:

* The subject must not have a history of anorexia nervosa.
* The subject must not have a history of clinically significant cardiac disease, any clinically significant abnormal cardiac condition, or be known to have a clinically significantly abnormal ECG. Specifically excluded conditions include coronary artery disease, clinically significant cardiac arrhythmias, and congestive heart failure.
* The subject must not have a history of stroke.
* The subject must not have a history of narrow angle glaucoma.
* The subject must not have an organic cause of obesity (e.g., untreated hypothyroidism).
* The subject must not have a history of seizures.
* The subject must not have severe renal or hepatic dysfunction.
* The subject must not be using any of the following medications while taking study medication: monoamine oxidase inhibitors (e.g., furazolidone, phenelzine, procarbazine HCl, selegiline), lithium, serotonin reuptake inhibitors, opioids (e.g., dextromethorphan, meperidine, pentazocine, fentanyl), prescribed or over-the-counter weight loss agents, centrally acting appetite suppressants, tryptophan, migraine agents (e.g., sumatriptan succinate, dihydroergotamine) or any other medication that, in the opinion of the Investigator, may pose harm to the subject, obscure the effects of study medication or interfere with the process of drug absorption, distribution, metabolism, or excretion (i.e., enzyme inducers or enzyme inhibitors). The regular use of sympathomimetics (e.g. cough and cold remedies, asthma medication) is contraindicated during the study. Study medication should be discontinued for 3 days before the use of opioids. THE SUBJECT SHOULD NOT BE TAKEN OFF ANTIDEPRESSANTS IN ORDER TO BE PLACED IN THE STUDY.
* The subject must not have a history of hypersensitivity to MERIDIA.
* The subject must not have a history of alcohol or drug addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 1998-09; Primary Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Body Weight Loss | Mean Change From Baseline

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Mean Change From Baseline
Waist/Hip Circumference | Mean Change From Baseline